CLINICAL TRIAL: NCT05206695
Title: The SIP Study: Simultaneously Implementing Pathways for Improving Asthma, Pneumonia, and Bronchiolitis Care for Hospitalized Children
Brief Title: Simultaneously Implementing Pathways for Improving Asthma, Pneumonia, and Bronchiolitis Care for Hospitalized Children
Acronym: SIP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Society of Hospital Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: R61HL157804 (NIH); R61HL157804 (NIH)
Record Dates: First submitted 2022-01-11; First posted 2022-01-25 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Asthma; Pneumonia; Bronchiolitis
Keywords: Children; Clinical pathways; Hospital
MeSH Terms: conditions — Asthma; Pneumonia; Bronchiolitis

STUDY DESIGN:
Intervention Model Description: Participating hospitals will be randomized into either an intervention group (will test simultaneous implementation of 3 clinical pathways) or control (will continue to provide standard care)
Who Masked: Outcomes Assessor
Masking Description: Participants, care providers, and investigators cannot be masked due to the nature of the intervention. However, outcomes assessors will be masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multi-condition Pathway Intervention (Experimental): The multi-condition pathway intervention consists of pathways clinicians select from to guide the care of children with asthma, pneumonia, or bronchiolitis. Key implementation strategies include audit and feedback, plan-do-study-act cycles, and electronic order sets.
  Interventions: Behavioral: Multi-condition Pathway Intervention
- Standard of Care (No Intervention): Hospitals randomized to the control arm will not receive the multi-condition pathway intervention or any external supports for implementation. They will continue to provide current standards of care.

INTERVENTIONS:
Behavioral: Multi-condition Pathway Intervention — See Experimental/Arm 1 description
  Arms: Multi-condition Pathway Intervention

SUMMARY:
This study's objective is to identify and test pragmatic and sustainable strategies for implementing a multi-condition clinical pathway intervention for children hospitalized with asthma, pneumonia, or bronchiolitis in community hospitals. The hypothesis is that the multi-condition pathway intervention will be associated with significantly greater increases in clinicians' adoption of evidence-based practices compared to control. The study is a pragmatic, cluster-randomized trial in US community hospitals. The primary outcome will be adoption of evidence-based practices over a sustained period of 2 years. Secondary outcomes include length of hospital stay, intensive care unit transfer, and hospital readmission/emergency department revisit.

DETAILED DESCRIPTION:
Asthma, pneumonia, and bronchiolitis are the top causes of childhood hospitalization in the US, leading to approximately 350,000 hospitalizations and $2 billion in costs annually. Poor guideline adoption by clinicians contributes to poor health outcomes for children hospitalized with these respiratory illnesses, including longer recovery time/hospital stay, higher rates of transfer to intensive care units, and increased risk of hospital readmission.

Pathways can improve clinicians' adoption of evidence-based practices/guidelines in both children's and community hospital settings. Pathways are simple, visual diagrams that guide clinicians step-by-step through the evidence-based care of a specific medical condition (accessed via paper or electronically). Most hospitals implement pathways for a single medical condition at a time (e.g., asthma). But Seattle Children's Hospital developed an intervention for simultaneously implementing pathways for multiple conditions. This intervention led to sustained guideline adoption, decreased length of stay, and decreased costs; and, these effects were comparable to those shown with single-condition pathway implementation. This multi-condition pathway intervention has not yet been studied in community hospitals, which face unique implementation barriers.

The study's objective is to identify and test pragmatic and sustainable strategies for implementing a multi-condition pathway intervention for children hospitalized with asthma, pneumonia, or bronchiolitis in community hospitals. The study is a pragmatic, cluster-randomized trial in US community hospitals. The pathway intervention will be implemented using the key implementation strategies defined for this intervention (audit and feedback, electronic health record integration, plan-do-study-act cycles). The primary outcome will be adoption of evidence-based practices over a sustained period of 2 years. Secondary outcomes include length of hospital stay, intensive care unit transfer, and hospital readmission/emergency department revisit.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of asthma AND age >2 to <18 years-old at time of admission to the hospital OR
* Primary diagnosis of pneumonia AND age >2 months and <18 years at time of admission to the hospital OR
* Primary diagnosis of bronchiolitis AND age <2 years at time of admission to the hospital

Exclusion Criteria:

* Diagnosis of SARS-CoV-2
* Transfer in from another inpatient facility
* Pre-existing chronic illnesses (e.g., lung disease, cardiovascular disease, neurologic disorders)

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 3840 (Estimated)
Dates: Start 2022-05-13 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Pneumonia Evidence Based Practice 1 | During a hospitalization, approximately 2 days
  Administration of narrow spectrum antibiotic
Pneumonia Evidence Based Practice 2 | During a hospitalization, approximately 2 days
  No prescription of macrolide antibiotics
Asthma Evidence Based Practice 1 | During a hospitalization, approximately 2 days
  Prescription of inhaled corticosteroids for children greater than or equal to 5 years-old
Asthma Evidence Based Practice 2 | During a hospitalization, approximately 2 days
  Use of metered-dose inhalers
Asthma Evidence Based Practice 3 | During a hospitalization, approximately 2 days
  Use of an asthma pathway/bronchodilator weaning protocol
Bronchiolitis Evidence Based Practice 1 | During a hospitalization, approximately 2 days
  No administration of bronchodilators
Bronchiolitis Evidence Based Practice 2 | During a hospitalization, approximately 2 days
  No chest radiographs

SECONDARY OUTCOMES:
Length of Hospital Stay | During a hospitalization, approximately 2 days
  Length Hospital Stay
Transfer to Intensive Care | During a hospitalization, approximately 2 days
  The event of patient being transferred to an ICU
30-day Hospital Readmission or Emergency Department Revisit | 30 days after hospital discharge
  Event of a patient being readmitted to hospital or having an emergency department visit within 30 days of hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Sunitha V Kaiser, MD, MSc, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Data generated under this project will be administered in accordance with the policies of the University of California San Francisco (UCSF) and NIH/NHLBI. The Final Research Data (the dataset necessary to document and support research findings) will be made available for sharing after the main research findings from the final data set have been accepted for publication in a peer-reviewed journal. Prior to sharing, data will be redacted to strip all direct identifiers of hospitals (no identifiers of patients/individuals will be collected).
Supporting Information: Study Protocol, SAP
Time Frame: The data will become available after peer-reviewed publication, and it will be available for 3 years.

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-09-11): https://cdn.clinicaltrials.gov/large-docs/95/NCT05206695/Prot_SAP_ICF_001.pdf